CLINICAL TRIAL: NCT05109052
Title: A Phase 1b/2 Trial of PXS-5505 Combined With First Line Atezolizumab Plus Bevacizumab For Treating Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Trial of PXS-5505 Combined With First Line Atezolizumab Plus Bevacizumab For Treating Patients With Unresectable Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no accrual of eligible participants
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nabeel Badri, Senior Instructor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGIH21023
Record Dates: First submitted 2021-09-15; First posted 2021-11-05 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma; Cancer of Liver
Keywords: Hepatocellular Carcinoma; Cancer of Liver; PXS-5505
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Open label safety and tolerability assessment of PXS-5505:
  (PXS-5505) 100-200mg BID (Atezolizumab) 1200mg every 3 weeks (Bevacizumab) 15mg/kg every 3 weeks
  Interventions: Drug: PXS-5505 and Atezolizumab and Bevacizumab

INTERVENTIONS:
Drug: PXS-5505 and Atezolizumab and Bevacizumab — Open label safety and tolerability assessment of PXS-5505 incorporating first-line combination therapy Atezolizumab and Bevacizumab

SUMMARY:
This trial will assess the safety and tolerability of PXS-5505 incorporating first-line combination therapy Atezolizumab and Bevacizumab in unresectable or metastatic hepatocellular carcinoma. Phase 2 will assess the efficacy of this combination therapy in unresectable or metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
Primary liver malignancies have doubled in incidence over the last two decades. These malignancies are now the 4th leading cause of cancer-related mortality worldwide with a 19.6% 5-year relative survival. Hepatocellular carcinoma (HCC) accounts for 90% with cholangiocarcinoma (CCA) accounting for the remainder. Currently, just 20-30% are resectable at presentation with many patients relying on systemic therapy. Beyond resection, effective systemic therapies are lacking, thus new treatment regimens are of significant clinical need. Recent phase III data with combination of Atezolizumab (anti-PD-L1) and Bevacizumab (anti-VEGF) as first-line therapy in unresectable HCC demonstrated improved progression-free and overall survival compared to Sorafenib, thus bringing immunotherapy to the forefront of combating this disease. Despite this improvement, patients experience significantly more adverse events with the addition of anti-VEGF therapy. This combination of Atezolizumab and Bevacizumab is an attractive immunotherapeutic backbone for pairing HCC therapy with means to improve drug delivery and boost response in order to decrease anti-VEGF dosing.

HCC most often develops in the background of chronic inflammation from sustained liver damage, hepatocyte cell death, and compensatory proliferation. During liver injury, hepatic stellate cells (HSCs) transform from quiescent to activated cells, characterized by altered matrix protease activity and deposition of extracellular matrix (ECM) proteins. ECM deposition increases liver stiffness that leads to vascular resistance and hypoxia, stimulating pro-angiogenic factors and subsequent angiogenesis. Secretion of growth factors (TGF-β, PDGF, and FGF-2) by the ECM and tumor cells, attracts fibroblasts from neighboring tissues and aids in transformation to cancer-associated fibroblasts (CAFs).[23] CAFs interplay with the ECM, contributing to further desmoplasia and remodeling through secretion of lysyl oxidases that catalyze collagen cross-linking. The accumulation of collagen cross-links results in marked increase in stromal stiffening and interstitial fluid pressure (IFP) reducing delivery of chemotherapy and immunotherapy Lysyl oxidases (LOX) are a family of 5 secreted copper-dependent amine oxidases (LOX, LOXL1-4) that catalyze the cross-linking of collagen and elastin in the extracellular matrix. High LOX expression has been show to correlate with poor prognosis across a variety of solid malignancies, including hepatocellular carcinoma. This trial pairs PXS-5505 (pan-lysyl oxidase inhibitor) with Atezolizumab and Bevacizumab in patients with unresectable or metastatic HCC. Phase 1b of this study will be an open label safety and tolerability assessment of PXS-5505 (pan-lysyl oxidase inhibitor) with a dose escalation design. The Phase 2 portion of the study will assess the efficacy of combination PXS-5505 with Atezolizumab and Bevacizumab compared to historical standard of care Atezolizumab and Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative must be able to understand and willing to sign an IRB approved written informed consent document.
* Patients must be 18 years or older
* Patient must have histological or radiographically confirmed unresectable or metastatic hepatocellular carcinoma.
* Patients must have no concomitant active oncologic diagnosis
* Patient must have at least one radiographically measurable lesion defined as non-radiated lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 10mm with calipers by radiographic exam. Further details listed in section 5.5.
* Patient must have received no previous systemic or investigational therapy for the treatment of HCC. Patients who previously received locoregional therapies remain eligible for this study.
* Patient must have a life expectancy of minimum 3 months.
* Patient must have normal bone marrow and organ function as defined below.

  * Absolute neutrophil count >1,500/mcl
  * Platelets >75,000/ul without transfusion
  * Hemoglobin >9.0 g/dL
  * Creatinine should be below the upper limit of normal OR
  * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Aspartate aminotransferase (AST), Alanine transaminase (ALT), and alkaline phosphatase (ALP) <5 times the upper limit of normal
  * Serum bilirubin no greater than 1.5-2x the upper limit of normal
* Patient not on anticoagulation must have international Normalized Ratio (INR) and activated partial thromboplastin time (PTT) <1.7 upper limit of normal. Patients on anticoagulation may be included, provided they can be off anticoagulation as indicated for paired biopsy collection.
* Patient will have an ECOG performance status of 0 or 1
* Patient must consent for baseline and on treatment biopsies, if prior baseline biopsies have been performed, and stored within the University of Rochester Cancer Library, then baseline biopsies are not necessary.
* Patients must be Child-Pugh class A or less
* Female subjects of childbearing potential must demonstrate a negative urine or serum pregnancy test.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) for a duration consistent with that described in the Bevacizumab and Atezolizumab labels (i.e. 6 months). Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Male subjects with a female partner of child-bearing potential must agree to use 2 adequate methods of contraception (barrier + hormonal for example).

Exclusion Criteria:

* Patient with any histologic variant of HCC such as fibrolamellar, sarcomatous, or mixed cholangiocarcinoma and HCC.
* Patient has a history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or prostate cancer that does not require treatment.
* Patient who received a previous systemic therapy for hepatocellular carcinoma or has tumor recurrence sooner than 6 months after completion of the last dose of therapy.
* Patient who is receiving any other investigational agent
* Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXS-5505, Atezolizumab, or Bevacizumab
* Patient with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, any clinically active malabsorption syndrome, inflammatory bowel disease, any condition that increases the risk of severe gastrointestinal toxicity, or psychiatric illness/social situations that would limit compliance with study requirements
* Has current active autoimmune disease, or a documented history of autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, resolved childhood asthma/atopy, hypothyroidism on thyroid supplementation, and type 1 diabetics would be exception to this rule.
* Patients who are eligible for liver transplantation
* Has had an allogenic tissue/solid organ transplant.
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
* Has received or plans to receive a live vaccine within 30 days prior to the first administration of study medication. Flu vaccines that do not contain live virus are permitted.
* Has known active Hepatitis B or C.
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Inadequately controlled arterial hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Evidence of bleeding diathesis or significant coagulopathy
* Inability to tolerate oral medications
* Child Pugh B or C cirrhosis
* Known connective tissue disorder
* Evidence of vascular aneurysmal disease
* History of myeloproliferative, myelodysplastic disorders, or monoclonal gammopathy of undetermined significance
* Major surgery within 4 weeks of enrollment
* Patient who is pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 10 years
  measured by adverse event severity and quantity

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Badri, Principal Investigator — Univ. of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided